CLINICAL TRIAL: NCT00833183
Title: A Study of Safety and Efficacy of Topical Methylaminolevulinate 80mg/g With and Without Occlusion Followed by Red Light Exposure in Subjects With Facial Acne
Brief Title: Safety and Efficacy Study of Topical Methyaminlevulinate (MAL) in Subjects With Facial Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Photocure (Industry)
Responsible Party: Per Fuglerud, Photocure
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INNO-6005
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 25 J/cm2, with occlusion on right side (Active Comparator): Subjects will receive MAL cream in a thin layer on both sides of the face (except nose and peri-ocular area) at a concentration of 80 mg/g). Occlusion will be applied to one half of the face. After an incubation time of 90 minutes both sides of the face will be exposed to either 25 J/cm2 of red light starting with the occluded side first.
  Interventions: Drug: MAL
- 37 J/cm2, with occlusion on right side (Active Comparator): Subjects will receive MAL cream in a thin layer on both sides of the face (except nose and peri-ocular area) at a concentration of 80 mg/g). Occlusion will be applied to one half of the face. After an incubation time of 90 minutes both sides of the face will be exposed to 37 J/cm2 of red light starting with the occluded side first.
  Interventions: Drug: MAL
- 25 J/cm2 , with occlusion on left side (Active Comparator): Subjects will receive MAL cream in a thin layer on both sides of the face (except nose and peri-ocular area) at a concentration of 80 mg/g). Occlusion will be applied to one half of the face. After an incubation time of 90 minutes both sides of the face will be exposed to either 25 J/cm2 of red light starting with the occluded side first.
  Interventions: Drug: MAL
- 37 J/cm2 , with occlusion on left side (Active Comparator): Subjects will receive MAL cream in a thin layer on both sides of the face (except nose and peri-ocular area) at a concentration of 80 mg/g). Occlusion will be applied to one half of the face. After an incubation time of 90 minutes both sides of the face will be exposed to 37 J/cm2 of red light starting with the occluded side first.
  Interventions: Drug: MAL

INTERVENTIONS:
Drug: MAL — 80 mg/g cream one administration with incubation for 90 minutes

SUMMARY:
A study of safety and efficacy of topical methyaminlevulinate 80mg/g with and without occlusion followed by red light exposure in subjects with facial acne.

DETAILED DESCRIPTION:
Photocure ASA has developed a cream formulation containing methyl aminolevulinate (MAL), an ester of ALA. There is extensive experience with the safety of MAL-PDT in humans.

This study will assess safety and efficacy of four treatments with methylaminolevulinate (MAL) at 80 mg/g performed with and without occlusion and followed by red light exposure 90 minutes later in subjects with facial acne vulgaris. Subjects will be randomized to one of two groups of 20 subjects: Group 1 will receive 25 J/cm2 of red light (45 mW/cm2) and group 2 will receive 37 J/cm2 of red light (90 mW/cm2). For each subject one side of the face will be randomized to receive MAL for 90 minutes without occlusion and the other side of the face will receive MAL for 90 minutes with occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Subject willing to use an adequate contraceptive method or is surgically sterile, post menopausal, abstinent or with a same-sex partner. Adequate means of contraception include; IUD in use 30 days prior to day 0, barrier methods and spermicide in use atleast 14 days prior to day 0 or oral contraceptive in use for at least 6 months prior to day 0
* Age 18 or older
* Capable of giving informed consent
* Diagnosis of acne vulgaris on the face with at least 10 inflammatory lesions on both sides of the face at screening and day 0
* Global acne severity assessment score ≥ 3 at the screening and day 0 visit.

Exclusion Criteria:

* Allergy to methylaminolevulinate or any component of the vehicle
* Acne fulminans or conglobata on the face
* Clinical significant sensitivity to visible light, porphyria or porphyrin sensitivity
* Use of any topical treatment for acne on the face within the previous 2 weeks before day 0
* Any use of systemic antibiotics within 1 month prior to day 0 or use of isotretinoin within 1 year prior to Day 0
* Exposure to ultraviolet radiation (UVB phototherapy, sun tanning salons) within 4 weeks of Day 0
* Use of any investigational drug within 4 weeks of Day 0
* Alcoholism or drug abuse in the past year
* Any unstable or serious medical condition at the discretion of the investigator
* Current pregnancy or lactation
* Use of hormonal contraceptives solely for control of acne
* Current use of oral contraceptives (unless subject is on a stable dose e.i. at least six months of treatment prior Day 0), testosterone or any other systemic hormonal treatment
* Any serious dermatological disorder, including malignancies that would either put the subject at risk or interfere with efficacy or safety evaluations
* Fitzpatrick phototype V or VI (inadequate penetration of red light in dark skin subjects)
* Subjects with extensive facial hair (e.g. beard) that would either impair red light exposure or interfere with lesion evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To compare the number of inflammatory acne lesions according to time on the side with occlusion and the side without occlusion for subjects with facial acne vulgaris exposed to 25 J/cm2 and 37 J/cm2 of red light. | 4 and 12 weeks after last PDT session.

SECONDARY OUTCOMES:
Exposed to 25 J/cm2 and 37 J/cm2 of red light and with and withut occlusion :-Compare number of non-inflammatory acne lesions. -Safety assesment of MAL-PDT. -Evaluate PAP photobleaching. | At each treatment visit and 2 and 7 days after first PDT treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD MSC FRCPC, Principal Investigator — Innovaderm Research Inc.
Locations (2):
- Canada (2):
  - Innovaderm Research Inc, Laval, Quebec
  - Innovaderm Research Inc., Montreal, Quebec